CLINICAL TRIAL: NCT04570098
Title: Prevalence and Prognostic Relevance of Tricuspid Regurgitation in Different Heart Failure Entities
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Henryk Dreger, Professor, Charite University, Berlin, Germany
Other Study IDs: EA1/178/19
Record Dates: First submitted 2020-09-20; First posted 2020-09-30 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Tricuspid Regurgitation; Heart Failure
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The present study includes patients with tricuspid regurgitation and heart failure diagnosed with echocardiography. The aim is to evaluate the physical performance of patients with tricuspid regurgitation and heart failure, to observe the course of the diseases and to allow a better understanding of new therapy options.

DETAILED DESCRIPTION:
Moderate to severe tricuspid regurgitation (TR) is a frequent result of left heart failure causing a limiting prognosis. The new interventional therapies have given more relevance to the questions of the prognostic significance of severe TR in the various heart failure entities.

Important but currently unanswered questions for the establishment of successful, interventional therapies of TR are:

1. What effect does TR have on patients with heart failure?
2. Which patients at which stage of the disease benefit from interventional TR-therapies? In order to answer these questions, the aim of the study is to prospectively record the prevalence of TR (including quantification) in all heart failure patients at the Charité, followed by long-term observation to assess its prognostic relevance.

In addition to answering the above-mentioned questions, the project will allow a central registration of all symptomatic heart failure patients. A comparative outcome analysis per propensity score matching with the untreated patients of the registry would allow to give first considerations which patients are ideal candidates for interventional therapies.

Primary endpoint: death Secondary endpoint: hospitalization due to cardiac decompensation, exercise capacity according to NYHA classification

ELIGIBILITY:
Inclusion Criteria:

* Patients with transthoracic echocardiography (TTE) and heart failure
* Reported heart failure symptoms within the last two years
* >18 years
* Written, documented consent

Exclusion Criteria:

- Patients in care or unable to consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population include patients with heart failure (all three entities). All patients will be examined with an echocardiography at the Charité, followed by long-term observation to assess the prognostic relevance of tricuspid regurgitation in heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 1016 (Actual)
Dates: Start 2020-07-26 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 3 months after enrolment
  Overall mortality after 3 months (number of deceased patients)
Overall mortality | 24 months after enrolment
  Overall mortality after 24 months (number of deceased patients)

SECONDARY OUTCOMES:
hospitalization due to cardiac decompensation | 3 months after enrolment
  number of hospitalized patients after 3 months
exercise capacity according to NYHA classification | 3 months after enrolment
hospitalization due to cardiac decompensation | 24 months after enrolment
  number of hospitalized patients after 24 months
exercise capacity according to NYHA classification | 24 months after enrolment

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
As part of the expected publications, it is planned to provide data of the study participants and more detailed information on inclusion and exclusion criteria (study protocol).